CLINICAL TRIAL: NCT00407615
Title: A DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED STUDY ON MAGNETIC FIELD THERAPY TO IMPROVE CHRONIC LUMBAR PAIN
Brief Title: Double-Blind Placebo Study on Magnetic Field Therapy in Chronic Lumbar Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Collaborators: Steven P. Cole, PhD. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12106
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Chronic Low Back Pain

INTERVENTIONS:
Device: Flex Pad/Static Magnet

SUMMARY:
This project is to assess the effectiveness of the use of magnets in reducing chronic lumbar pain. I understand that I will wear a flex pad (magnet) during waking hours and keep daily Visual Analog Scale (VAS) pain scores to determine if wearing this device will reduce my constant pain. I understand that there are no adverse side effects known from the use of these magnets other than irritation at the site. The identical inactive pads (sham/placebo) have been supplied for use as controls.

I will be randomly assigned into one of two groups and I agree to remain blinded as to the specific type of device that I will receive, i.e. active vs. placebo. Dr. Weintraub (principal investigator) will remain blinded throughout the study. I also agree to not break the blind. Dr. Weintraub has stated that as a result of my cooperation and ability to complete the study, I will be guaranteed to either keep my specific device or receive a specific known "active" device gratis. This currently sells commercially for $60.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this study is to determine if treatment with a flex pad impregnated with static/permanent magnets that can penetrate over 70 mm may improve the quality of chronic lumbar pain with reduction of pain scores.

HYPOTHESIS:

It is my hypothesis that the application of a flex pad active magnetic therapy vs. sham if utilized daily during waking hours can reduce back pain and/or radicular pain. The null hypothesis is that treatment of subjects with chronic back pain with exposure to static/permanent magnetic fields have no measurable effect on chronic back pain scores and will be equal to the underlying placebo.

SIGNIFICANCE:

This is a low-cost, safe and effective, non-invasive treatment for musculoskeletal pain and specifically for chronic low back pain. An effective outcome would reduce dependency on pharmacological interventions with attempt at reductions in known side effects.

DESIGN:

This is a double-blind, randomized, placebo-controlled study which will consist of two treatment groups. Treated subjects will receive a static/permanent magnetic flex pad with a nominal strength of less than 1000 Gauss. Control subjects will receive physically identical flex pad without magnet with a nominal surface field strength of 0 Gauss (placebo). The magnets will be contained in a pad with a Velcro cover and subjects will wear the pad attached to their undergarments/skin during waking hours. Dr. Weintraub will examine participants initially to look for presence or absence of radiculitis, range of motion, presence of absence of spasm, etc. The primary outcome measures will be reduction of chronic low back pain in comparison with prior baseline scores. It is recognized that these changes are subjective in nature. Patients will maintain their VAS scores on a monthly basis and at the end of the study, individuals will return all forms and be reevaluated by Dr. Weintraub. They will be asked specific questions regarding PGIC for bias, etc.

PARTICIPANTS:

Forty (40) outpatients with chronic low back pain will be enrolled.

PROTOCOL:

A DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED STUDY ON MAGNETIC FIELD THERAPY TO IMPROVE CHRONIC LUMBAR PAIN

INCLUSION CRITERIA:

* Female or male subjects age 18-80.
* Capable of understanding and complying with study protocols.
* Chronic lumbar pain for at least six months.

EXCLUSION CRITERIA:

* Unable to understand informed consent (mental retardation, psychosis, communicative impairment).
* Cardiac pacemaker or other mechanical internal devices.
* Tumor in the spine/history of malignancy or tumor.
* Pregnancy.
* Prior spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain

Exclusion Criteria:

* No surgery on spine,
* no tumor,
* no pacemaker,
* no pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-12; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures will be reduction of chronic low back pain in comparison with prior baseline scores

CONTACTS AND LOCATIONS:
Overall Officials: Steve P Cole, PhD, Study Chair — Research Design Inc.
Locations (2):
- United States (2):
  - Dr. Michael I. Weintraub, Briarcliff, New York
  - Michael I. Weintraub MD 325 S. Highland Avenue, Briarcliff, New York